CLINICAL TRIAL: NCT00355511
Title: Heart Failure Evaluation Acute Referral Team Trial (HEARTT)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit patients
Sponsor: University of Alberta (Other)
Responsible Party: Dr. Ross Tsuyuki, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPICORE2006-002
Record Dates: First submitted 2006-07-18; First posted 2006-07-24 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Heart Failure, Congestive
Keywords: heart failure, congestive; patient care team; randomized controlled trial; disease management; drug therapy; diet therapy; hospitalization; mortality
MeSH Terms: conditions — Heart Failure | interventions — Dosage Forms; Self Care; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: education: disease, medication, self-care, diet — education on heart failure self care; medication initiation and titration, frequent follow-up

SUMMARY:
The purpose of this study is to assess the impact of a multidisciplinary team clinic including a clinical pharmacist, a registered nurse (RN), dietician and physician providing short-term sub-acute management of patients with heart failure on patient outcomes and the quality of medication use. Patients being discharged from the emergency department with a diagnosis of heart failure will be eligible for this study. We believe that emergency room visits, hospitalization and deaths secondary to heart failure will decrease secondary to this program.

DETAILED DESCRIPTION:
BACKGROUND: Heart failure (HF)accounts for morbidity and mortality in Canada. In contrast to coronary heart disease, the mortality rate attributed to HF has decreased minimally, only 14%, over the last 35 years. This is despite a plethora of new therapeutic modalities proven to decrease mortality in HF. HF is also one of the leading causes of hospitalizations accounting for the second highest total number of hospital days and the third highest number of patients affected. It has been estimated that approximately 20-50% of patients will be readmitted to hospital with one year. Patients seen in the emergency department (ED)and discharged home from the ED are also at high risk for readmissions. A local study by our group indicated that 44% of patients seen for HF in the ED have this disposition and as such have a strikingly 50% higher readmission rate at 30 days compared to those admitted to hospital. This difference could be explained by a "care gap" as evidence by a low utilization of both angiotensin converting enzyme inhibitors and beta-blockers in this group. However, a lack of patient education on self-care and follow-up post ED discharge could also attribute to these rates. We propose testing a intervention employing a multidisciplinary team to facilitate follow-up, provide HF education, including self-care, and improve utilization of proven drug-therapy in patients discharged with HF from the ED on the outcomes of hospitalizations and mortality.

PURPOSE: To improve the quality of care for patient with HF

HYPOTHESIS: Multidisciplinary team management of patients with HF has be shown to decrease both morbidity and mortality in HF patients. A multifaceted program including rapid referral, early short-term follow-up, medication initiation and titration and HF education in collaboration with a dietician, nurse, pharmacist and physician will improve HF patient care in terms of clinical outcomes, quality of life and evidence-based medication utilization.

STUDY DESIGN: The study will utilize an unblinded randomized controlled trial (RCT) design. Eligible patients will included patient discharged from the ED with a diagnosis of heart failure. All patients referred from the ED will be seen in a rapid referral clinic within 1 week. Eligible patients will then randomized to an intervention arm or usual care. The usual care group will have a consultation letter with recommendations sent their family doctor and will receive a booklet on heart failure. The intervention arm will be followed in clinic monthly by the multidisciplinary team. Medication will be initiated and titrated to target dose. Patients will receive education regarding heart failure, medications, lifestyle, diet and self-management. Communication will the patient's primary care provider will also be enhanced.

SIGNIFICANCE: The literature describes a plethora of therapeutic modalities aimed at improving the care of patients with HF. However, in terms of multifaceted disease management interventions, the majority of HF studies have examined high risk patients that were admitted to hospital or stable outpatients. This proposed study would examine a unique population of patients being discharged from the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency department (ED) with signs and symptoms of heart failure with a plan to discharge home from the ED .

Exclusion Criteria:

* < 18 years of age
* planned follow-up with Cardiology or Internal Medicine post discharge from ED
* heart transplant candidate or recipient
* current Heart Function Clinic patient
* left ventricular ejection fraction >0.40
* unable or unwilling to attend clinic visits
* heart failure requiring admission to hospital
* patients living outside the Capital Health catchment area
* participation in another heart failure clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Difference in the composite endpoint of emergency room visits, hospitalizations, and mortality at 6 months between the intervention and usual care group. | 6 months

SECONDARY OUTCOMES:
Difference in the following between the intervention and usual care groups at 6 months: emergency room visits, hospitalizations, mortality, proportion of patients utilizing evidence-based therapies, quality of life | 6 months
Description of the implementation of the rapid assessment clinic | 6 months
Patient satisfaction | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ross T Tsuyuki, PharmD, MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- See also: Related Info — https://www.epicore.ualberta.ca